CLINICAL TRIAL: NCT04648540
Title: Multimodal Opioid-free Anesthesia Versus Opioid-based Anesthesia for Patients Undergoing Cardiac Valve Surgeries: A Randomized Controlled Trial
Brief Title: Multimodal Opioid-free Anesthesia Versus Opioid-based Anesthesia for Patients Undergoing Cardiac Valve Surgeries: RCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hossam El-Ashmawi, Professor of anesthiology and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD-242-2019
Record Dates: First submitted 2020-11-04; First posted 2020-12-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine; Pregabalin; Acetaminophen; Ketorolac; Celecoxib; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Free Anesthesia (OFA) (Experimental): The following drugs will be administered 10 minutes before induction of anesthesia in group I (OFA):
  * Pregabalin 150 mg orally with a small sip of water
  * Acetaminophen 1 gm and Ketorolac 30 mg in 100 mL i.v. over 10 minutes
  * Dexmedetomidine loading dose of 0.5 mic/kg i.v. over 10 minutes
  * Lidocaine loading dose of 1.5 mg/kg i.v. over 10 minutes
  For simplicity, the weight-based doses of dexmedetomidine and lidocaine will be prepared in a 20 mL syringe
  the following drugs will be administered as a continuous infusion:
  * Dexmedetomidine 0.5 mic/kg/h
  * Lidocaine 0.5 mg/kg/h
  Patients in both groups will be extubated when they meet our institutional criteria for extubation. Postoperative analgesia will be started as follows:
  Group I (OFA):
  * Acetaminophen 1 gm/6h
  * ketorolac 30 mg/8h
  * Pregabalin 150 mg once at night
  * Celecoxib 200 mg/24 hours
  Interventions: Drug: Dexmedetomidine 0.5 mic/kg/h
- Opioid Anesthesia (OA) (Active Comparator): Before induction In Group II (OA) patients will receive placebo pills and normal saline in equivalent volumes .
  Maintenance
  In Group II (OA) patients will receive a continuous infusion of Fentanyl (1 mic/kg/h)
  Patients in both groups will be extubated when they meet our institutional criteria for extubation. Postoperative analgesia will be started as follows:
  • Morphine 0.1 mg /kg PRN every 8 hours
  Interventions: Drug: Fentanyl 1 mic/kg/hr

INTERVENTIONS:
Drug: Dexmedetomidine 0.5 mic/kg/h — In Group I (OFA) the following drugs will be administered preoperatively:
  Acetaminophen 1 gm and Ketorolac 30 mg in 100 mL i.v. over 10 minutes Dexmedetomidine loading dose of 0.5 mic/kg i.v. over 10 minutes Lidocaine loading dose of 1.5 mg/kg i.v. over 10 minutes
  The following drugs will be administered as a continuous infusion throughout the operation:
  * Dexmedetomidine 0.5 mic/kg/h
  * Lidocaine 0.5 mg/kg/h
  The following drugs will be administered postoperatively:
  Acetaminophen 1 gm/6h ketorolac 30 mg/8h Pregabalin 150 mg once at night Celecoxib 200 mg/24 hours
  Other Names: Lidocaine 0.5 mg/kg/h; Pregabalin 150 mg; Acetaminophen 1g; Ketorolac 30 mg; Celecoxib 200 mg
  Arms: Opioid-Free Anesthesia (OFA)
Drug: Fentanyl 1 mic/kg/hr — In Group II (OA) patients will receive a continuous infusion of Fentanyl (1 mic/kg/h) Morphine 0.1 mg/kg PRN will be administered every 8 hours for postoperative analgesia
  Other Names: Morphine 0.1 mg/kg/hr
  Arms: Opioid Anesthesia (OA)

SUMMARY:
Several studies demonstrated the effectiveness of OFA in patients undergoing non-cardiac surgery. Preoperative use of Cox inhibitors, GABA analogues and acetaminophen have been shown to decrease use of opioids postoperatively . Intraoperative use of agents that lead to opioid sparing effects via sodium channel blockade, blockade of G protein-coupled receptors, NMDA blockade, central alpha-2 agonists and anti-inflammatory effects can make opioid-free anesthesia (OFA) possible. On the other hand, there have been no studies demonstrating the effectiveness of an OFA technique in patients undergoing cardiac surgery except for two case reports who successfully implemented the OFA regimen in two patients undergoing valve replacement surgeries. The investigators therefore propose this prospective randomized controlled trial to investigate whether a multimodal opioid-free anesthesia regimen will be suitable as an alternative to conventional opioid-based regimen in patients undergoing valve surgery

DETAILED DESCRIPTION:
High-dose opioid anesthesia during cardiac surgery has been the mainstay of cardiac anesthesia for decades due to its ability to preserve hemodynamic stability and attenuate hormonal and metabolic response to surgical stress (1) . However, large doses of long-acting opioids required patients to be ventilated post-operatively for 12-24 h. Modifications in these practices have been dictated by the increasing cost, complications of prolonged mechanical ventilation, and the changes in demographics of patients presenting for cardiac surgery (2) . Moreover, the intraoperative use of large bolus doses or continuous infusions of potent opioids may be associated with postoperative hyperalgesia and tolerance (3). When it comes to ambulatory surgery, opioid related side effects, such as postoperative nausea and vomiting (PONV), prolonged sedation, ileus and urinary retention may delay recovery and discharge or cause unanticipated hospital readmission (4) . Such complications might, at least in part, also apply to cardiac anesthesia.

Recent evidence suggests that increased total dose of opioids during cardiac surgery may lead to increased in-hospital, as well as long-term post-operative pain medication requirements for up to one year (5). Moreover, according to Hirji et al study , ongoing opioid use three months after CABG was present in 21.7% of opioid-exposed patients versus 3.2% of opioid-naive patients (6). In addition, Opioids have many known side effects such as somnolence, brainstem and respiratory depression , and chronic opioid dependence (7-9), and there is a national trend to decrease opioid use during non-cardiac surgery to promote faster recovery and decrease narcotic use post-operatively (1) .

Several studies demonstrated the effectiveness of Opioid-free Anesthesia (OFA) in patients undergoing non-cardiac surgery(4,10,11). Preoperative use of COX inhibitors, GABA analogues and acetaminophen have been shown to decrease use of opioids postoperatively(10). Intraoperative use of agents that lead to opioid sparing effects via sodium channel blockade, blockade of G protein-coupled receptors, NMDA blockade, central alpha-2 agonists and anti-inflammatory effects can make opioid-free anesthesia (OFA) possible (12,13). On the other hand, there have been no studies demonstrating the effectiveness of an OFA technique in patients undergoing cardiac surgery except for two case reports who successfully implemented the OFA regimen in two patients undergoing valve replacement surgeries (14,15). The investigators therefore propose this prospective randomized controlled trial to investigate whether a multimodal opioid-free anesthesia regimen will be suitable as an alternative to conventional opioid-based regimen in patients undergoing valve surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiac valve surgeries ( replacement or repair ) .
2. Age (18-80) years
3. Both sexes

Exclusion Criteria:

* Patient refusal
* Known allergy to any of the medications used in the study
* Combined valve and CABG surgeries
* Redo surgery
* Infective endocarditis
* Patients in heart failure or heart block or with significant systolic dysfunction (EF < 40%) or diastolic dysfunction more than grade II
* Pregnant females
* Patients being treated for chronic pain or with recent use (< two weeks) of opioids, gabapentin, or pregabalin.
* Substance abuse
* Patients with renal impairment (creatinine > 2 mg/dL) or hepatic impairment (ALT > 2 folds, INR > 1.5 and/or serum albumin < 2.5 g/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Extubation time (min) | 24 hours
  Extubation time, defined as the time from discontinuation of inhalation agents to extubation

SECONDARY OUTCOMES:
Heart rate (beats/min) | 24 hours
  HR
  o Arterial blood pressure (systolic, diastolic, and mean)
Blood pressure (mm Hg) | 24 hours
  Systolic, diastolic, and mean blood pressure
Postoperative rescue analgesia (number) | 24
  The number of patients requiring rescue analgesia with Morphine
Postoperative morphine consumption (mg) | 24 hours
  The total dose of morphine administered

CONTACTS AND LOCATIONS:
Overall Officials: hossam El-Ashmawi, Professor, Principal Investigator — Cairo University
Locations (1):
- Kasr Al Ainy School of Medicine Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Rong LQ, Kamel MK, Rahouma M, Naik A, Mehta K, Abouarab AA, Di Franco A, Demetres M, Mustapich TL, Fitzgerald MM, Pryor KO, Gaudino M. High-dose versus low-dose opioid anesthesia in adult cardiac surgery: A meta-analysis. J Clin Anesth. 2019 Nov;57:57-62. doi: 10.1016/j.jclinane.2019.03.009. Epub 2019 Mar 11. PMID 30870677
- [Background] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Background] Lavand'homme P, Steyaert A. Opioid-free anesthesia opioid side effects: Tolerance and hyperalgesia. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):487-498. doi: 10.1016/j.bpa.2017.05.003. Epub 2017 May 17. PMID 29739537
- [Background] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031
- [Background] van Gulik L, Ahlers SJ, van de Garde EM, Bruins P, van Boven WJ, Tibboel D, van Dongen EP, Knibbe CA. Remifentanil during cardiac surgery is associated with chronic thoracic pain 1 yr after sternotomy. Br J Anaesth. 2012 Oct;109(4):616-22. doi: 10.1093/bja/aes247. Epub 2012 Jul 24. PMID 22831889
- [Background] Hirji SA, Landino S, Cote C, Lee J, Orhurhu V, Shah RM, McGurk S, Kaneko T, Shekar P, Pelletier MP. Chronic opioid use after coronary bypass surgery. J Card Surg. 2019 Feb;34(2):67-73. doi: 10.1111/jocs.13981. Epub 2019 Jan 9. PMID 30625257
- [Background] Macintyre PE, Walker SM. The scientific evidence for acute pain treatment. Curr Opin Anaesthesiol. 2010 Oct;23(5):623-8. doi: 10.1097/ACO.0b013e32833c33ed. PMID 20811175
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Alam A, Juurlink DN. The prescription opioid epidemic: an overview for anesthesiologists. Can J Anaesth. 2016 Jan;63(1):61-8. doi: 10.1007/s12630-015-0520-y. Epub 2015 Oct 27. PMID 26507535
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] James MF. Magnesium: an emerging drug in anaesthesia. Br J Anaesth. 2009 Oct;103(4):465-7. doi: 10.1093/bja/aep242. No abstract available. PMID 19749114
- [Background] Landry E, Burns S, Pelletier MP, Muehlschlegel JD. A Successful Opioid-Free Anesthetic in a Patient Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2517-2520. doi: 10.1053/j.jvca.2018.11.040. Epub 2018 Nov 28. No abstract available. PMID 30611614
- [Background] Cardinale JP, Gilly G. Opiate-Free Tricuspid Valve Replacement: Case Report. Semin Cardiothorac Vasc Anesth. 2018 Dec;22(4):407-413. doi: 10.1177/1089253218771342. Epub 2018 Apr 20. PMID 29676223
- [Background] Salah M, Hosny H, Salah M, Saad H. Impact of immediate versus delayed tracheal extubation on length of ICU stay of cardiac surgical patients, a randomized trial. Heart Lung Vessel. 2015;7(4):311-9. PMID 26811837